CLINICAL TRIAL: NCT03159650
Title: Randomized Comparative Study Between Intravascular Ultrasonography Guided and Angiography-guided Recanalization of Coronary Chronic Total Occlusions
Brief Title: Comparative Study Between Intravascular Ultrasonography Guided and Angiography-guided Recanalization of Coronary Chronic Total Occlusions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Osman Abdelhamead, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: IVUSAN
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Coronary Occlusion
MeSH Terms: conditions — Coronary Occlusion | interventions — Ultrasonography, Interventional

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravascular ultrasonography guided (Experimental)
  Interventions: Device: intravascular ultrasonography
- Angiography guided (Active Comparator)
  Interventions: Device: intravascular ultrasonography

INTERVENTIONS:
Device: intravascular ultrasonography — intravascular ultrasonography will be used during the study for the resolving proximal cap ambiguity of chronic total occlusion, facilitating re-entry into the true lumen after subintimal crossing and confirming distal true lumen guidewire position

SUMMARY:
Chronic total occlusion is defined as thrombolysis in myocardial infarction (TIMI) flow grade 0 with an estimated duration of at least 3 months. The interest in chronic total occlusion (CTO) percutaneous coronary intervention (PCI) has increased, but with failure rate up to 20%, leading to important developments in dedicated equipment and techniques.

In the 2014 European Guidelines on Myocardial Revascularization, intravascular ultrasound was recommended to guide stent implantation in selected patients, and this recommendation was a class IIa/level of evidence B.

In CTO PCI, certain angiographic features such as blunt proximal CTO cap, tortuosity, heavy calcification, and lack of visibility of path in the distal vessel increase procedural difficulty

ELIGIBILITY:
Inclusion Criteria:

* patients with coronary angiography showing chronic coronary total

Exclusion Criteria:

1. Acute coronary syndrome within 3 months.
2. Patients with previous coronary artery bypass graft (CABG).
3. Patients with known renal insufficiency (eGFR < 60 ml/kg/m2, serum creatinine ≥ 2.5 mg/dL, or on dialysis).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
outcomes of intravascular ultrasound guided re-canalized CTO during the procedure and composite of cardiac death, myocardial infarction, or target vessel revascularization | 6 months
  the study will assess the composite of cardiac death, myocardial infarction, or target vessel revascularization, rehospitalization, coronary artery bypass surgery and stroke within both groups

REFERENCES:
- [Background] Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Uva MS, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A; Grupa Robocza Europejskiego Towarzystwa Kardiologicznego (ESC); Europejskie Stowarzyszenie Chirurgii Serca i Klatki Piersiowej (EACTS) do spraw rewaskularyzacji miesnia sercowego; European Association for Percutaneous Cardiovascular Interventions (EAPCI). [2014 ESC/EACTS Guidelines on myocardial revascularization]. Kardiol Pol. 2014;72(12):1253-379. doi: 10.5603/KP.2014.0224. No abstract available. Polish. PMID 25524605
- [Background] Park Y, Park HS, Jang GL, Lee DY, Lee H, Lee JH, Kang HJ, Yang DH, Cho Y, Chae SC, Jun JE, Park WH. Intravascular ultrasound guided recanalization of stumpless chronic total occlusion. Int J Cardiol. 2011 Apr 14;148(2):174-8. doi: 10.1016/j.ijcard.2009.10.052. Epub 2009 Nov 26. PMID 19942305
- [Background] Stone GW, Reifart NJ, Moussa I, Hoye A, Cox DA, Colombo A, Baim DS, Teirstein PS, Strauss BH, Selmon M, Mintz GS, Katoh O, Mitsudo K, Suzuki T, Tamai H, Grube E, Cannon LA, Kandzari DE, Reisman M, Schwartz RS, Bailey S, Dangas G, Mehran R, Abizaid A, Moses JW, Leon MB, Serruys PW. Percutaneous recanalization of chronically occluded coronary arteries: a consensus document: part II. Circulation. 2005 Oct 18;112(16):2530-7. doi: 10.1161/CIRCULATIONAHA.105.583716. No abstract available. PMID 16230504